CLINICAL TRIAL: NCT03185013
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of VGX-3100 Delivered Intramuscularly Followed by Electroporation With CELLECTRA™-5PSP for the Treatment of HPV-16 and/or HPV-18 Related High Grade Squamous Intraepithelial Lesion (HSIL) of the Cervix
Brief Title: REVEAL 1 (Evaluation of VGX-3100 and Electroporation for the Treatment of Cervical HSIL)
Acronym: REVEAL 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPV-301; 2016-002761-63 (EudraCT Number)
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cervical Dysplasia; Cervical High Grade Squamous Intraepithelial Lesion; HSIL
Keywords: Cervical intraepithelial neoplasia (CIN); Human papillomavirus (HPV); High grade squamous intraepithelial lesion (HSIL); CIN 2; CIN 3; papillomavirus
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions | interventions — VGX-3100; Electroporation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- VGX-3100 + EP (Experimental): Participants received three IM injections of 6 milligram (mg) (in 1 milliliter [mL]) VGX-3100 followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
  Interventions: Biological: VGX-3100; Device: Electroporation (EP)
- Placebo + EP (Placebo Comparator): Participants received three IM injections of 1 mL VGX-3100 matching placebo followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
  Interventions: Biological: Placebo; Device: Electroporation (EP)

INTERVENTIONS:
Biological: VGX-3100 — 1 mL VGX-3100 will be injected IM and delivered by EP using CELLECTRA™-5PSP on Day 0, Week 4 and Week 12.
  Arms: VGX-3100 + EP
Biological: Placebo — 1 mL of Placebo will be injected IM and delivered by EP using CELLECTRA™-5PSP on Day 0, Week 4 and Week 12.
  Arms: Placebo + EP
Device: Electroporation (EP) — Intramuscular injection followed by EP with the CELLECTRA™ 5PSP device.

SUMMARY:
HPV-301 is a prospective, randomized, double-blind, placebo controlled Phase 3 study to determine the efficacy, safety, and tolerability of VGX-3100 administered by intramuscular (IM) injection followed by electroporation (EP) delivered with CELLECTRA™ 5PSP in adult women with histologically confirmed cervical high grade squamous intraepithelial lesion (HSIL) (cervical intraepithelial neoplasia grade 2 [CIN2] or grade 3 [CIN3]) associated with human papillomavirus (HPV) 16 and/or HPV-18.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and above
* Confirmed cervical infection with HPV types 16 and/or 18 at screening
* Cervical tissue specimen/slides provided to Study Pathology Adjudication Committee for diagnosis scheduled to be collected within 10 weeks prior to anticipated date of first dose of study drug
* Confirmed histologic evidence of cervical HSIL at screening
* Must be judged by Investigator to be an appropriate candidate for the protocol-specified procedure required at Week 36
* With respect to their reproductive capacity must be post-menopausal or surgically sterile or willing to use a contraceptive method with failure rate of less than 1% per year when used consistently and correctly from screening until Week 36
* Normal screening electrocardiogram (ECG)

Exclusion Criteria:

* Microscopic or gross evidence of adenocarcinoma-in-situ (AIS), high grade vulvar, vaginal, or anal intraepithelial neoplasia or invasive cancer in any histopathologic specimen at screening
* Cervical lesion(s) that cannot be fully visualized on colposcopy
* History of endocervical curettage (ECC) which showed cervical HSIL indeterminate, or insufficient for diagnosis
* Treatment for cervical HSIL within 4 weeks prior to screening
* Pregnant, breastfeeding or considering becoming pregnant during the study
* History of previous therapeutic HPV vaccination
* Immunosuppression as a result of underlying illness or treatment
* Receipt of any non-study, non-live vaccine within 2 weeks of Day 0
* Receipt of any non-study, live vaccine within 4 weeks of Day 0
* Current or history of clinically significant, medically unstable disease or condition which, in the judgment of the investigator, would jeopardize the safety of the participant, interfere with study assessments or endpoint evaluation, or otherwise impact the validity of the study results
* Presence of acute or chronic bleeding or clotting disorder that would contraindicate IM injections, or use of blood thinners within 2 weeks of Day 0
* Participation in an interventional study with an investigational compound or device within 30 days of signing informed consent
* Less than two acceptable sites available for IM injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (60):
- United States (22):
  - Mesa Obstetricians and Gynecologist, Mesa, Arizona
  - Women's Health Research, Scottsdale, Arizona
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Women's Medical Research Group, Clearwater, Florida
  - Altus Research, Lake Worth, Florida
  - Salom and Tangir LLC, Miramar, Florida
  - Comprehensive Clinical Trials LLC, West Palm Beach, Florida
  - Augusta University, Augusta, Georgia
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Saginaw Valley Medical Research Group LLC, Saginaw, Michigan
  - Meridian Clinical Research Norfolk, Norfolk, Nebraska
  - New Jersey Medical School, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Suffolk Obstetrics and Gynecology, Port Jefferson, New York
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Greenville Pharmaceutical Research, Inc., Greenville, South Carolina
  - Magnolia Ob/Gyn Research Center, LLC, Myrtle Beach, South Carolina
  - Chattanooga Medical Research Inc, Chattanooga, Tennessee
  - Women's Physician Group, Memphis, Tennessee
  - UAG Innovation Women Research, LLC, Houston, Texas
  - Group For Women, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
- Argentina (3):
  - Instituto de Ginecología, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía
- Belgium (2):
  - Centre Hospitalier Universitaire Ambroise Paré, Mons, Hainaut
  - Ziekenhuis Oost-Limburg, Genk, Limburg
- Estonia (3):
  - Pärnu Hospital, Pärnu, Pärnumaa
  - East Tallinn Central Hospital Womens Clinic, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Kätilöopiston sairaala, Helsinki
  - Lääkäriasema Cantti Oy, Kuopio
- Germany (2):
  - Elisabeth Krankenhaus Essen GmbH, Essen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Italy (3):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale Dei Tumori, Milan
- Lithuania (2):
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - Vilnius District Central Outpatient Clinic, Vilnius
- Nuevo Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco, Mexico
- Peru (2):
  - Unidad de Ensayos Clinicos (UNIDEC) del Policlinico Universidad Nacional Mayor de San Marcos, Lima
  - Liga Peruana De Lucha Contra El Cancer, Lima
- Perpetual Succour Hospital, Cebu, Philippines
- Poland (3):
  - Niepubliczny Zakład Opieki Zdrowotnej Profimed, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin, Lublin Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice
- Portugal (2):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
- Puerto Rico Translational Research Center (PRTRC), Rio Piedras, Puerto Rico
- Slovakia (2):
  - MCM GYNPED, s.r.o., Dubnica nad Váhom
  - Univerzitna nemocnica Martin, Martin
- South Africa (2):
  - Lynette Reynders Private Practice, Centurion, Gauteng
  - University of Cape Town, Cape Town
- Spain (3):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Thailand (2):
  - Chulalongkorn University, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
- United Kingdom (2):
  - Aberdeen Royal Infirmary - PPDS, Aberdeen
  - St Marys Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 96 study centers in 20 countries from 28 June 2017 to 6 April 2021.
Pre-assignment Details: A total of 201 participants with human papillomavirus (HPV)-16 and/or HPV-18 related high-grade squamous intraepithelial lesion (HSIL) of the cervix were randomized in this study, 138 in VGX-3100+EP and 63 in Placebo + EP.
Groups:
- VGX-3100 + Electroporation (EP): Participants received three IM injections of 6 milligram (mg) (in 1 milliliter [mL]) VGX-3100 followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
Period: Overall Study
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Started | 138 | 63
Intent-to-Treat (ITT) Population (ITT population included all participants who were randomized.) | 138 | 63
Modified ITT (mITT) Population (mITT population included all participants who received at least one dose of clinical trial treatment and who had the analysis endpoint of interest.) | 134 | 63
Safety Population (Safety set included all participants who received at least one dose of clinical trial treatment.) | 136 | 63
Completed | 116 | 56
Not Completed | 22 | 7
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Progressive Disease | 1 | 0
Not completed — Lost to Follow-up | 8 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Deviation | 2 | 0
Not completed — Reason not Specified | 3 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who were randomized.
Groups:
- VGX-3100 + Electroporation (EP): Participants received three IM injections of 6 mg (in 1 mL) VGX-3100 followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
- Total: Total of all reporting groups
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP | Total
Number analyzed (Participants) | 138 | 63 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (6.53) | 31.9 (6.08) | 31.5 (6.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 63 | 201
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 9 | 31
  Not Hispanic or Latino | 112 | 54 | 166
  Unknown or Not Reported | 4 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 6 | 15
  Black or African American | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 109 | 46 | 155
  Other | 10 | 2 | 12
  Multiple | 1 | 0 | 1
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Evidence of Cervical HSIL on Histology and No Evidence of HPV-16 and/or HPV-18 in Cervical Samples
Description: Participants with no histologic (i.e., biopsies or excisional treatment) evidence of cervical HSIL, no evidence of HPV-16 and/or HPV-18 at the Week 36 time frame, and participants in which excision or biopsy sample was not obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined by histology as negative, squamous atypia, or low-grade intraepithelial lesion (LSIL). Cervical samples for HPV-16 and/or HPV-18 were collected using the ThinPrep®.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 22.5 | 11.1
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the one-sided p-value was <0.025 and the corresponding lower bound of the 95% CI exceeded zero (0); p = 0.029, Miettinen and Nurminen method; Difference in percentage = 11.4, 95% CI 2-sided [-0.4 to 21.2]

2. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs) Following Investigational Treatment for the Duration of the Study
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. An SAE is any experience that suggested a significant hazard, contraindication, side effect, or precaution, and fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: From baseline up to Week 88
Population: Safety set included all participants who received at least one dose of clinical trial treatment. One participant received mixed treatment and was excluded from the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 136 | 62
Participants
  Number of Participants with any AE | 131 | 61
  Number of Participants with any SAE | 13 | 6

3. Secondary Outcome: Percentage of Participants With No Evidence of Cervical HSIL on Histology
Description: Participants with no histologic (i.e., biopsies or excisional treatment) evidence of cervical HSIL at Week 36 and participants in which an excision or biopsy sample was not obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 31.9 | 19.0
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in percentage = 12.8, 95% CI 2-sided [-0.6 to 24.5]

4. Secondary Outcome: Percentage of Participants With No Evidence of HPV-16 and/or HPV-18 in Cervical Samples by Type Specific HPV Testing
Description: Participants with no evidence of HPV-16 and/or HPV-18 at the Week 36 time frame and participants in which an excision or biopsy sample was not obtained between the initial dose up to Week 36 were considered to be responders. Cervical samples for HPV-16 and/or HPV-18 were collected using the ThinPrep®.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 34.1 | 15.9
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in percentage = 18.2, 95% CI 2-sided [5.1 to 29.4]

5. Secondary Outcome: Percentage of Participants With No Evidence of LSIL or HSIL on Histology
Description: Participants with no histologic evidence of cervical HSIL, squamous atypia, or LSIL at the Week 36 time frame and participants in which an excision or biopsy sample was not obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined as no evidence of cervical squamous intraepithelial neoplasia 1 (CIN1), CIN2, or CIN3 on biopsies or excisional treatment.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 24.6 | 11.1
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in percentage = 13.5, 95% CI 2-sided [1.7 to 23.5]

6. Secondary Outcome: Percentage of Participants With No Evidence of LSIL or HSIL and No Evidence of HPV-16 and/or HPV-18
Description: Participants with no histologic evidence of cervical HSIL, squamous atypia, and LSIL, no evidence of HPV-16 and/or HPV-18 by type specific HPV testing at the Week 36 time, and participants in which an excision or biopsy sample was not obtained between initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined as no evidence of CIN1, CIN2, or CIN3 on biopsies or excisional treatment.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 18.1 | 6.3
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in percentage = 11.8, 95% CI 2-sided [1.5 to 20.3]

7. Secondary Outcome: Percentage of Participants With No Progression of Cervical HSIL to Cervical Carcinoma
Description: Participants with no histologic evidence of cervical Adenocarcinoma in situ or cervical carcinoma at the Week 36 timeframe relative to baseline and participants in which an excision or biopsy sample was not obtained between initial dose up to Week 36 were considered as responders.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 84.1 | 85.7
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in percentage = -1.7, 95% CI 2-sided [-11.5 to 10.3]

8. Secondary Outcome: Percentage of Participants Who Have Cleared HPV-16 and/or HPV-18 in Non-cervical Anatomic Locations
Description: Participants with no evidence of HPV-16 and/or HPV-18 on specimens from noncervical anatomic locations (oropharynx, vagina and intra-anal) at the Week 36 time frame were considered as responder.
Time Frame: Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 138 | 63
percentage of participants | 20.3 | 9.5
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in percentage = 10.8, 95% CI 2-sided [-0.5 to 20.1]

9. Secondary Outcome: Levels of Serum Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations
Description: A standardized binding enzyme-linked immunosorbent assay (ELISA) was performed to measure the anti-HPV-16/18 antibody response induced by VGX-3100.
Time Frame: Week 15 and Week 36
Population: mITT population included all participants who received at least one dose of clinical trial treatment and who had the analysis endpoint of interest. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Median (Full Range); unit: reciprocal endpoint titer
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 128 | 61
reciprocal endpoint titer
  HPV-16 E7 at Week 15 | 225.0 [1 to 18225] | 1.0 [1 to 6075]
  HPV-16 E7 at Week 36: number analyzed (Participants) | 128 | 58
  HPV-16 E7 at Week 36 | 1.0 [1 to 18225] | 1.0 [1 to 6075]
  HPV-18 E7 at Week 15 | 2025.0 [1 to 18225] | 1.0 [1 to 18225]
  HPV-18 E7 at Week 36: number analyzed (Participants) | 128 | 58
  HPV-18 E7 at Week 36 | 225.0 [1 to 18225] | 1.0 [1 to 2025]
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Week 15: HPV-16 E7; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Location shift = 224.0, 95% CI 2-sided [24.0 to 224.0]
Statistical Analysis 2: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Week 36: HPV-16 E7; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Location shift = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 3: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Week 15: HPV-18 E7; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Location Shift = 2024.0, 95% CI 2-sided [2000.0 to 6050.0]
Statistical Analysis 4: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Week 36: HPV-18 E7; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Location Shift = 224.0, 95% CI 2-sided [74.0 to 674.0]

10. Secondary Outcome: Change From Baseline in Interferon-Gamma Response Magnitude
Description: Assessment of cellular immune activity occurred via the application of the Interferon-γ enzyme-linked immunosorbent spot (IFN-γ ELISpot). Peripheral blood mononuclear cells (PBMCs) isolated from whole blood sample were used for analysis.
Time Frame: Baseline; Week 15 and Week 36
Population: as for outcome 9
Measure: Median (Full Range); unit: spot forming units (SFU)/10^6 PBMC
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 116 | 54
spot forming units (SFU)/10^6 PBMC
  HPV-16 E6: Baseline | 0.83 [0.0 to 40.0] | 0.00 [0.0 to 16.7]
  HPV-16 E6: Change from Baseline at Week 15: number analyzed (Participants) | 102 | 45
  HPV-16 E6: Change from Baseline at Week 15 | 13.33 [0.0 to 446.7] | 0.00 [0.0 to 13.3]
  HPV-16 E6: Change from Baseline at Week 36: number analyzed (Participants) | 90 | 41
  HPV-16 E6: Change from Baseline at Week 36 | 8.33 [0.0 to 780.0] | 0.00 [0.0 to 25.0]
  HPV-16 E7: Baseline | 0.00 [0.0 to 53.3] | 0.00 [0.0 to 83.3]
  HPV-16 E7: Change from Baseline at Week 15: number analyzed (Participants) | 102 | 45
  HPV-16 E7: Change from Baseline at Week 15 | 10.83 [0.0 to 213.3] | 0.00 [0.0 to 13.3]
  HPV-16 E7: Change from Baseline at Week 36: number analyzed (Participants) | 90 | 41
  HPV-16 E7: Change from Baseline at Week 36 | 7.50 [0.0 to 81.7] | 0.00 [0.0 to 8.3]
  HPV-18 E6: Baseline | 0.00 [0.0 to 10.0] | 0.00 [0.0 to 20.0]
  HPV-18 E6: Change from Baseline at Week 15: number analyzed (Participants) | 102 | 45
  HPV-18 E6: Change from Baseline at Week 15 | 50.83 [0.0 to 1910.0] | 0.00 [0.0 to 6.7]
  HPV-18 E6: Change from Baseline at Week 36: number analyzed (Participants) | 90 | 41
  HPV-18 E6: Change from Baseline at Week 36 | 38.33 [0.0 to 1031.7] | 0.0 [0.0 to 23.3]
  HPV-18 E7: Baseline | 0.00 [0.0 to 11.7] | 0.00 [0.0 to 91.7]
  HPV-18 E7: Change from Baseline at Week 15: number analyzed (Participants) | 102 | 45
  HPV-18 E7: Change from Baseline at Week 15 | 14.17 [0.0 to 251.7] | 0.00 [0.0 to 20.0]
  HPV-18 E7: Change from Baseline at Week 36: number analyzed (Participants) | 90 | 41
  HPV-18 E7: Change from Baseline at Week 36 | 10.00 [0.0 to 508.3] | 0.00 [0.0 to 6.7]
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-16 E6: Week 15; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Location shift = 11.67, 95% CI 2-sided [8.33 to 20.00]
Statistical Analysis 2: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-16 E6: Week 36; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 8.33, 95% CI 2-sided [3.33 to 11.67]
Statistical Analysis 3: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-16 E7: Week 15; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 10.83, 95% CI 2-sided [5.00 to 15.00]
Statistical Analysis 4: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-16 E7: Week 36; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 7.50, 95% CI 2-sided [1.67 to 10.00]
Statistical Analysis 5: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-18 E6: Week 15; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 50.83, 95% CI 2-sided [31.67 to 66.67]
Statistical Analysis 6: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-18 E6: Week 36; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 38.33, 95% CI 2-sided [18.33 to 51.67]
Statistical Analysis 7: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-18 E7: Week 15; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 14.17, 95% CI 2-sided [6.67 to 18.33]
Statistical Analysis 8: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; HPV-18 E7: Week 36; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 10.00, 95% CI 2-sided [5.00 to 15.00]

11. Secondary Outcome: Change From Baseline in Flow Cytometry Response Magnitude
Description: Assessment of cellular immune activity was measured using the application flow cytometry for the purposes of performing a Lytic Granule Loading Assay. The Lytic Granule Loading assay examines the following external cellular markers: CD3, CD4, CD8 (T cell identification), CD137, CD38 and CD69 (T cell activation markers) as well as PD-1 (exhaustion/activation marker). Here change from baseline in CD8+CD137+Perforin+, CD8+CD38+Perforin+ and CD8+CD69+Perforin+ are reported.
Time Frame: Baseline, Week 15
Population: as for outcome 9
Measure: Median (Full Range); unit: SFU/10^6 PBMC
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
Number analyzed (Participants) | 114 | 58
SFU/10^6 PBMC
  CD8+CD137+Perforin+: Baseline: number analyzed (Participants) | 114 | 48
  CD8+CD137+Perforin+: Baseline | 0.004 [0.00 to 0.15] | 0.001 [0.00 to 0.22]
  CD8+CD137+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 106 | 42
  CD8+CD137+Perforin+: Change from Baseline at Week 15 | 0.035 [0.00 to 0.44] | 0.000 [0.00 to 0.10]
  CD8+CD38+Perforin+: Baseline: number analyzed (Participants) | 114 | 48
  CD8+CD38+Perforin+: Baseline | 0.000 [0.00 to 0.21] | 0.000 [0.00 to 0.12]
  CD8+CD38+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 106 | 42
  CD8+CD38+Perforin+: Change from Baseline at Week 15 | 0.011 [0.00 to 0.23] | 0.000 [0.00 to 0.10]
  CD8+CD69+Perforin+: Baseline: number analyzed (Participants) | 114 | 48
  CD8+CD69+Perforin+: Baseline | 0.009 [0.00 to 0.11] | 0.001 [0.00 to 0.13]
  CD8+CD69+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 106 | 42
  CD8+CD69+Perforin+: Change from Baseline at Week 15 | 0.044 [0.00 to 0.37] | 0.000 [0.00 to 0.07]
Statistical Analysis 1: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Parameter: CD8+CD137+Perforin+; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 0.025, 95% CI 2-sided [0.002 to 0.046]
Statistical Analysis 2: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Parameter: CD8+CD38+Perforin+; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 0.011, 95% CI 2-sided [0.000 to 0.014]
Statistical Analysis 3: Comparison: VGX-3100 + Electroporation (EP) vs Placebo + EP; Parameter: CD8+CD69+Perforin+; Test type: Superiority — Superiority was concluded if the lower bound of the 95% CI exceeded 0; Difference in median = 0.044, 95% CI 2-sided [0.017 to 0.058]

ADVERSE EVENTS:
Time Frame: From baseline up to Week 88
Description: Safety set included all participants who received at least one dose of clinical trial treatment. One participant received mixed treatment and was excluded from the safety analysis.
Arm/Group | VGX-3100 + Electroporation (EP) | Placebo + EP
All-Cause Mortality (participants affected / at risk) | 1/136 | 0/62
Serious Adverse Events (participants affected / at risk) | 13/136 | 6/62
Other Adverse Events (participants affected / at risk) | 131/136 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 + Electroporation (EP) (N=136) | Placebo + EP (N=62)
Adenosquamous Carcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Squamous Cell Carcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Diaphragmatic Hernia (Gastrointestinal disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 + Electroporation (EP) (N=136) | Placebo + EP (N=62)
Nausea (Gastrointestinal disorders) | 25 | 11
Abdominal Pain (Gastrointestinal disorders) | 8 | 4
Injection Site Pain (General disorders) | 105 | 49
Fatigue (General disorders) | 40 | 18
Injection Site Pruritus (General disorders) | 34 | 14
Injection Site Erythema (General disorders) | 33 | 14
Injection Site Swelling (General disorders) | 28 | 15
Injection Site Bruising (General disorders) | 14 | 9
Injection Site Haematoma (General disorders) | 8 | 6
Malaise (General disorders) | 9 | 5
Nasopharyngitis (Infections and infestations) | 13 | 4
Vaginitis Bacterial (Infections and infestations) | 9 | 4
Vulvovaginal Candidiasis (Infections and infestations) | 9 | 3
Urinary Tract Infection (Infections and infestations) | 7 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 6
Headache (Nervous system disorders) | 46 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03185013/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03185013/SAP_001.pdf